CLINICAL TRIAL: NCT05432973
Title: Efficacy of Percutaneous Electrical Nerve Stimulation Compared With Passive Assisted Neurodynamics in Brachial Plexus Neuropathy: a Pilot Randomized Controlled Trial.
Brief Title: Percutaneous Electrical Nerve Stimulation Compared to Passive Assisted Neurodynamics in Brachial Plexus Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PENS210722
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Percutaneous Electrical Nerve Stimulation; Peripheral Neuropathy; Neuropathic Pain
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neuralgia | interventions — Transcutaneous Electric Nerve Stimulation; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENS (Experimental)
  Interventions: Procedure: Percutaneous Electrical Nerve Stimulation
- Neurodynamics and manual therapy (Active Comparator)
  Interventions: Procedure: Neurodynamic and manual therapy

INTERVENTIONS:
Procedure: Percutaneous Electrical Nerve Stimulation — In the PENS treatment, a biphasic continuous waveform current with a frequency of 2 Hz, a pulse width of 50 microseconds and an intensity that produces visible motor responses of the innervated muscles was used, below the patient's pain threshold. The NT6021 Percutaneous Neuromodulation equipment of the Nutek® brand distributed by Fisiolab Ibérica® was used. This equipment has the CE marking, which denotes compliance with the requirements of the legislation of Royal Decree 414/1996 of March 1, which regulates medical devices. B.O.E. of April 24, 1996
  Arms: PENS
Procedure: Neurodynamic and manual therapy — The manual therapy consisted of passive-assisted mobilization and massage therapy of the muscular and fascial tissue, beginning with the cervical area, kneading while asking the patient to rotate the neck and then in the same way along the muscles and soft tissues innervated by the target nerve.
  Neurodynamic was performed in a passive-assisted manner, combining the patient's cervical mobilizations with the mobility of the upper limbs adapted to each case.
  Arms: Neurodynamics and manual therapy

SUMMARY:
Brachial plexus neuropathies, specifically of the median, radial, ulnar, suprascapular, axillary and dorsal scapular nerves, can arise when a peripheral nerve trunk or nerve root is subjected to injury, compression, inflammation or ischemia, resulting in reduced physical capabilities of the peripheral nervous system. Although pharmacological treatments provide mild symptomatic relief in the short term, they are not without side effects.

Neurostimulation techniques may be an effective treatment option for peripheral brachial plexus neuropathies. Some of these procedures are transcutaneous electrical nerve stimulation (TENS) or percutaneous electrical nerve stimulation (PENS). Although some case series have documented a positive effect in relation to ultrasound-guided PENS for subjects with subacromial pain syndrome or postsurgical pain, the lack of studies, to our knowledge, analyzing the effects of percutaneous electrical nerve stimulation, in relation to pain and paresthesias in subjects with brachial plexus neuropathy, warrants investigation for this goal.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with upper limb neural symptomatology between 18 and 60 years of age, presenting two or more of the following conditions:
* Paresthesias in any territory of the shoulder girdle, arm or hand
* Pain at rest in any territory of the upper extremity.
* Pain at rest in any upper extremity territory
* Sensations of electric shock in any territory of the shoulder girdle, arm or hand.
* Allodynia or cutaneous hyperalgesia in any territory of the shoulder girdle, arm or hand.

Exclusion Criteria:

* Less than 2 weeks of evolution
* Fracture in the affected upper extremity
* Suffering from another joint disorder such as osteoarthritis or rheumatic disease
* Suffering from generalized neuropathies due to neuromuscular disease or medication
* Inability to understand instructions or sign informed consent.
* Wearing a pacemaker or any electrical device implanted in the body
* Epilepsy
* Aversion or fear of needles
* Pregnant.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Lanss Scale | 10 minutes
  Useful to identify patients with a pain experience dominated by neuropathic mechanisms. It is based on the analysis of sensory description and exploration of sensory dysfunction at the patient's bedside. It consists of 7 items and is scored from 0 to 24. At a score of less than 12, the neuropathic component is considered unlikely. A score greater than or equal to 12 is considered probable neuropathic pain. It is a validated scale for patients with neuropathic pain.
Pain Detect Scale | 10 minutes
  Screening questionnaire for neuropathic pain. This scale consists of a section dedicated to pain intensity and another that is responsible for assessing the qualitative aspect of pain, i.e., identifying whether the pain is of neuropathic characteristics. In the total of this scale the maximum possible score is 38 points and the minimum -1. For screening purposes, a score less than or equal to 12 is considered an unlikely neuropathic component. A score greater than or equal to 19 concludes that the neurological component in pain is probable.
Numerical Pain Rating Scale (NPRS) | 1 minute
  A unique 11-point numerical scale validated in patients with various painful conditions. Data obtained through NPRS are easily documented, intuitively interpretable, and meet regulatory requirements for pain assessment and documentation. This scale is reliable and validated for assessing patients with pain20. Score 0 corresponds to "no pain" and score 10 corresponds to "maximum possible pain". In this study, patients were asked to mark their maximum pain detected in the last week (NPRS Max) and their minimum pain detected in the last week (NPRS Min).

SECONDARY OUTCOMES:
Neural stress test | 5 minutes
  Nerves react to certain mechanical stresses and forces, but to establish positivity of such tests, the possibilities of "false positivity" due to other non-nerve structures must first be eliminated. The determination of a positive neural test is established by provocation and symptom relief techniques. In this outcome measure only a positive or negative test was considered. The test was positive if the patient's neural symptoms were reproduced during provocation, or negative if no such symptoms occurred.
DASH scale | 5 minutes
  It is a validated scale for assessing upper limb functionality. It is an instrument that can be completed by the patient with the help of the physical therapist. It consists of 30 questions that assess certain symptoms, as well as the ability to perform activities, ranging from 1 to 5, with 1=no difficulty and 5=maximum difficulty. The higher the score, the greater the upper limb disability.
Thermography | 10 minutes
  A thermal camera, HT-02D infrared thermographic and visible light camera with IR 1024 pixels and -20~300°C, 6Hz refresh rate, infrared thermometer was used. The thermograph indicates the approximate temperature of the body segment to be examined by focusing it with the thermographic camera.

CONTACTS AND LOCATIONS:
Locations (1):
- Physiotherapy and exercise center Origenkinesis, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes